CLINICAL TRIAL: NCT02869100
Title: Comparison of Sodium Fluoride Positron Emission Tomography and Magnetic Resonance Imaging of Spine and Sacroiliac Joints for Detection of Inflammatory Lesions in Patients Affected by Spondyloarthritis
Brief Title: Comparison of Sodium Fluoride Positron Emission Tomography and Magnetic Resonance Imaging of Spine and Sacroiliac Joints for Detection of Inflammatory Lesions in Spondyloarthritis Patients
Acronym: FNa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-A00568-35
Record Dates: First submitted 2016-08-09; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Spondyloarthritis
Keywords: magnetic resonance imaging; sodium fluoride positron emission tomography
MeSH Terms: conditions — Spondylarthritis | interventions — Blood Specimen Collection; Magnetic Resonance Spectroscopy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Spondyloarthritis Patients (Experimental)
  Interventions: Other: Blood sample; Procedure: Sodium fluoride Positron Emission Tomography; Other: Magnetic Resonance Imaging; Other: Radiography

INTERVENTIONS:
Other: Blood sample
Procedure: Sodium fluoride Positron Emission Tomography
Other: Magnetic Resonance Imaging
Other: Radiography

SUMMARY:
The purpose is to compare detection of axial inflammatory lesions in patients affected by spondyloarthritis (SpA) with sodium fluoride positron emission tomography (PET) and magnetic resonance imaging (MRI), the reference technique.

It would be interesting to show the superiority of sodium fluoride PET on MRI for diagnosis of inflammatory lesions. It could be used for diagnostic care but also therapeutic care of patients with early forms of spondyloarthritis.

Secondary purposes are:

* To evaluate performances of sodium fluoride PET in detection of SpA peripheral damage (except spine and sacroiliac joints)
* To evaluate bone inflammation (axial and peripheral) with sodium fluoride PET and compare these data to clinic-biologic parameters used in clinical practice (BASDAI, BASFI, BASMI, sedimentation rate, C-reactive protein (CRP)) and to structural evaluation (sacroiliac New York, mSASSS and BASRI scoring methods)
* To study correlation of axial and peripheral bone inflammation (spine and sacroiliac joints) evaluated with sodium fluoride PET with biologic markers of inflammation and bone remodeling (MMP-3; DKK-1, IL-6, IL-17, TNF-α).

Known biologic markers of inflammation in SpA are correlated to activity obtained with MRI. It is interesting to compare to activity obtained with PET. Moreover, it has been recently showed the disassociation of inflammation and structural progression (anti-TNF treatments do not prevent structural progression) that is associated to markers of bone remodeling whose activity is influenced by an activation/inhibition system of biologic markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 year-old patients affected by axial or mixed SpA (ASAS criteria) or >18 year-old patients according to New York criteria
* Patients with bone marrow edema lesions in sacroiliac joints and/or spine detected with MRI
* No therapeutic changes between hospitalization for evaluation of SpA activity and inclusion visit
* Informed consent
* Affiliation to social security plan

Exclusion Criteria:

* Refusal or impossibility of signed informed consent
* Doubt about possible pregnancy in women of childbearing potential
* Pregnancy and breastfeeding
* History of drug addiction, alcoholism, psychological problems, severe co-morbidities
* Renal insufficiency (creatinine clearance < 60 ml/min)
* Juridical protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Concordance between binary topographic evaluations of bone inflammation in PET data and MRI data | up to 4 weeks
  presence or absence of inflammatory sites (MRI) or hyperfixation (PET) in 28 sites (24 vertebrae and 4 sacroiliac joints)
Concordance between semi-quantitative evaluation of bone inflammation in MRI data and PET data | up to 4 weeks
  PET: BME score adapted to PET for spine and modified SPARCC score adapted to PET for sacroiliac joints
  MRI: Berlin score BME for spine and SPARCC score for sacroiliac joints

SECONDARY OUTCOMES:
Structural evaluation with New York score | day 0
Structural evaluation with mSASSS scores | day 0
Structural evaluation with BASRI score | day 0
Levels of specific biologic markers of inflammation and bone remodeling in blood | up to 4 weeks
  MMP-3, DKK-1, IL-6, IL-17, TNF-α
Standard biologic evaluation of sedimentation rate | day 0
Standard biologic evaluation of C-reactive protein | day 0
Evaluation of spinal mobility with BASMI index | up to 4 weeks
Evaluation of disease activity with BASDAI index | up to 4 weeks
Evaluation of functional impact with BASFI index | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pierre OLIVIER, Pr, Principal Investigator — CHU de Nancy, Hôpitaux de Brabois, service de Médecine Nucléaire
Locations (1):
- CHU de Nancy, Hôpitaux de Brabois, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No